CLINICAL TRIAL: NCT01892137
Title: Histological Confirmation of Clinical Clearance of Actinic Keratoses Following Treatment With Ingenol Mebutate Gel, 0.05%
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP0041-62
Record Dates: First submitted 2013-06-23; First posted 2013-07-04 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2015-03

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; Histopathology; Reflectance Confocal Microscopy; Local Skin Reaction
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label active (Other)
  Interventions: Drug: Ingenol mebutate gel 0.05%

INTERVENTIONS:
Drug: Ingenol mebutate gel 0.05% — Once daily for 2 consecutive days

SUMMARY:
The main purpose of this trial is to demonstrate the predictive value of the clinical diagnosis of clearance of Actinic Keratoses after treatment with Ingenol Mebutate using histopathological examination as the standard.

ELIGIBILITY:
Inclusion Criteria:

* Must be male or female and at least 18 years of age.
* Female patients must be on non-childbearing potential or if of childbearing potential then negative serum and urine pregnancy test and using effective contraception
* Ability to provide informed consent
* Subjects must have 5-9 clinically typical, visible and discrete AK lesions within a contiguous 25cm2 treatment area on the trunk and extremities except the back of the hand
* AK should be confirmed by histopathology of one of the AK's prior to inclusion

Exclusion Criteria:

* location of the selected treatment area within 5cm of an incompletely healed wound or within 10cm of a suspected basal cell carcinoma or squamous cell carcinoma
* undergone Cosmetic or therapeutic procedures
* use of acid-containing therapeutic products within 2cm of the selected treatment area in the 2 weeks prior to Visit 1
* use of topical creams/lotions, artificial tanners or topical steroids within 2cm of the selected treatment areas in the 2 weeks prior to visit 1.
* treatment with immunomodulators, or interferon/interferon inducers or systemic medications that suppress the immune system within 4 weeks of visit 1
* treatment with 5-FU, imiquimod, diclofenac, ingenol mebutate of photodynamic therapy within 2cm of the treatment area in the 8 weeks prior to visit 1
* use of systemic retinoids
* those who are currently participating in any other interventional clinical trial
* females who are pregnant or are breastfeeding
* those known or suspected of not being able to comply with the requirements of the protocol or provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Clearance of AK | 8 weeks
  The primary response criterion is the clinical and histological clearance of AK at Day 57. Clinical Clearance will be measured by counting AKs, and histological clearance will be by performing a biopsy (result reported as AK or not AK).

SECONDARY OUTCOMES:
Complete clearance of AKs in the Selected Treatment Area | 8 weeks
  Efficacy in terms of complete clearance of AKs in the STA and histological clearance of pre-identified lesion. AK clearance will be determined by AK count. Clearance of the pre-identified lesion will be assessed by a histopatholgist from a biopsy sample and reported as AK or not AK.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Ulrich, Principal Investigator — Collegium Medicum Berlin GmbH, Germany
Locations (10):
- Australia (6):
  - Southderm Pty Ltd, Kogarah, New South Wales
  - Melanoma Institute Australia, North Sydney, New South Wales
  - The Skin Centre, Benowa, Queensland
  - South East Dermatology Centre, Carina Heights, Queensland
  - St John of God Dermatology, Subiaco, Western Australia
  - Burswood Dermatology, Victoria Park, Western Australia
- Germany (4):
  - Klinik für Dermatologie & Allergologie Klinikum Augsburg Süd, Augsburg
  - Collegium Medicum Berlin GmbH, Berlin
  - Medizinisches Zentrum Bonn Friedensplatz, Bonn
  - Hautarztpraxis Prof. Dr. med. C. Termeer, Stuttgart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: LEO Pharma — http://www.leopharma.com
- See also: Therapeutic Goods Administration — http://www.tga.gov.au
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en